CLINICAL TRIAL: NCT00702169
Title: Continuous Monitoring of the Lungs Ventilation Dynamics During Mechanical Ventilation by Small Surface Patches That Include Safe Motion Sensors
Brief Title: Continuous Monitoring of the Lungs Ventilation Dynamics During Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Dany Waisman, MD, Directon Newborn Unit, Carmel Medical Center
Other Study IDs: Neo- 01/2006
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Mechanical Ventilation
Keywords: high frequency ventilation monitoring; lung disease; Respiratory distress syndrome; lung barotrauma; mechanical ventilation; endotracheal tube displacement; endotracheal tube occlusion; one lung intubation
MeSH Terms: conditions — Lung Diseases; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Premature and term newborn infants (male/female)

SUMMARY:
Background: Patients that suffer from respiratory failure and need mechanical ventilation are at risk of further deterioration due to complications induced by progression of lung disease or the mechanical ventilation. The complications usually develop in a progressive manner, but are currently detected relatively late, when there is already severe and life threatening deterioration in patient oxygenation and sometimes irreversible damages.

Objective:To measure chest wall dynamics, derived from sensors placed on the chest and abdomen.

Methods: The system comprises of patches attached to the chest wall and upper abdomen that include mechanical sensors that measure the mechanics of lung inflation and deflation.

DETAILED DESCRIPTION:
Patients that suffer from respiratory failure and need mechanical ventilation are at risk of further life threatening deterioration following the development of mechanical problems related to airway management, development of lung barotrauma or displacement of the endotracheal tube.

Neonates especially need tight and sensitive monitoring of lung ventilation, because of the high prevalence of lung disease and need for ventilatory support in this population.

Methods:

The system comprises of patches attached to the chest wall and to the epigastrium. The patches include sensors that measure the mechanics of the lung inflation and deflation.

Study protocol

Following parental informed consent, three patches will be placed on both sides of the chest and over the epigastric area in infants that require tight respiratory monitoring.

The patches will be placed just beside the ECG patches. The placement of the patches will be performed by a physician. The monitoring can be preformed as long as the baby needs a tight respiratory monitoring. The patches will be replaced according to routine replacement policy of patches in the neonatal intensive care units, and at the regular time defined by the attending staff, and no longer than 24 hours. At the end of the data acquisition, the patches will be removed.

No additional intervention is required. The patient will be inspected by the supervising physician involve in the research.

It will not provide any data that may alter the treatment and will not interfere or influence the other monitoring devices that are used to evaluate the clinical status of the patient.

The other parameters that are regularly monitored, that are displayed on the bedside monitor and respirator will be recorded by the research assistant. The ventilated baby will be identified by a study number. There will be a separate database for the measurements and the demographic and clinical data. There will be no disclosure of the patient's identity along with the data analysis and publication of the results or communication to authorities or other medical practitioners.

Equipment safety:

The system is safe for the use in human subjects. The whole system is approved for safety according to the acquired standard ICE-60601

ELIGIBILITY:
Inclusion Criteria:

* Babies receiving respiratory support

Exclusion Criteria:

* Parental refusal to be included in the study
* Premature babies under 700 grams birth weight
* Prematurity below 26 weeks gestation
* Severe edematous babies (Hydrops fetalis)
* Severe Hypoxic Ischemic Encephalopathy, initial brain injury or severe intracranial bleeding or major congenital anomalies
* Skin reactions to the adhesive patches

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies receiving respiratory support, born at 26 weeks and over & birth weight 700 grams.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
A data-bank of measured changes in lung dynamics at various clinical settings acquired by the chest sensors.

SECONDARY OUTCOMES:
Detection of changes in lung ventilation by the novel system. Feasibility study. Comparison of the detection made by the novel system to the conventional monitoring methods in use.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Waisman, MD, Principal Investigator — Department of Neonatology Carmel Medical Center
Locations (1):
- Department of Neonatology, Carmel Medical Center, Haifa, Israel